CLINICAL TRIAL: NCT03122041
Title: Dipeptidyl Peptidase-4 (DPP-4) Inhibitor Sitagliptin Improved Beta Cell Function and Prevented a Conversion Rate to Impaired Glucose Tolerance IGT and Type 2 Diabetes T2D in Metformin Intolerant Obese Women With Polycystic Ovary Syndrome PCOS
Brief Title: Sitagliptin Improved Beta Cell Function and Prevented a Conversion Rate to Impaired Glucose Tolerance and Type 2 Diabetes in Metformin Intolerant Obese Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Simona Ferjan, MD, Principal Investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Metformin Intolerant PCOS
Record Dates: First submitted 2017-04-10; First posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: PCOS
Keywords: metformin intolerance; PCOS; Sitagliptin; beta cell function
MeSH Terms: interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SITA (Experimental): Sitagliptin (SITA) Lifestyle intervention and sitagliptin 100mg per day for 12 weeks
  Interventions: Drug: Sitagliptin; Behavioral: Lifestyle intervention
- CON (Experimental): Controls (CON) Lifestyle intervention
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Drug: Sitagliptin
  Other Names: Januvia
  Arms: SITA
Behavioral: Lifestyle intervention

SUMMARY:
Metformin is the first-line therapy for PCOS with high metabolic risk, yet a large proportion of patients cannot tolerate it due to associated gastrointestinal adverse events. The alternative pharmacological strategy when metformin cannot be tolerated is not well established in this population. Our aim was to evaluate whether sitagliptin (SITA) preserves metabolic profile in metformin (MET) intolerant PCOS with high metabolic risk.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old to menopause
* polycystic ovary syndrome (ASRM-ESHRE Rotterdam criteria)
* BMI of 30 kg/m2 or higher

Exclusion Criteria:

* significant cardiovascular disease
* significant kidney or hepatic disease
* personal or family history of medullary thyroid carcinoma
* known history of gallbladder disease
* known history of pancreatitis

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The main outcome was change in HOMA-β index (Homeostasis model assessment for beta cell function index). | Homeostasis model assessment for beta cell function index (HOMA-β) was calculated at the base point and after 12 weeks of clinical trial.

SECONDARY OUTCOMES:
The secondary outcome was change in fasting plasma glucose level (G0) | Patient's fasting glucose level was measured at the base point and after 12 weeks of clinical trial.
The secondary outcome was change in plasma glucose level at 120 minutes (G120) after glucose load in oral glucose tolerant test (OGTT). | Patient's plasma glucose level at 120 minutes (G120) after glucose load in oral glucose tolerant test (OGTT) was measured at the base point and after 12 weeks of clinical trial.

IPD SHARING:
Plan to Share IPD: No